CLINICAL TRIAL: NCT06396182
Title: Effect of Virtual Reality Exercise Versus Aerobic Training on Performance and Endurance in Physical Therapy Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Neama Mahmoud abd El-halim El-sheikh, physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004374
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cardiorespiratory Fitness or Endurance
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Group A (Study group): (Thirty participant) The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller).
  Group B (Control group): (Thirty participant) The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of cycling session by traditional stationary bike.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Study group): (Experimental): The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller).
  Interventions: Other: group (A ) study group :virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller).
- Group B (Control group): (Active Comparator): The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of cycling session by traditional stationary bike.
  - Cycling by traditional stationary bike: Participants will require to continuously pedal using the pulse oximeter for HR monitor. Research personnel monitored participants during the session adjusting pedal-resistance to ensure that the participants stayed within their target HR zone. (Daniel et al., 2020).
  Interventions: Other: group (A ) study group :virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller).

INTERVENTIONS:
Other: group (A ) study group :virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller). — group (A ) study group : virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller):
  The VR cycling session utilized the VZFIT VR Exercise Bike (VZFIT, Cambridge, MA), games were selected as preliminary pilot trials indicated these games to be most intense. Players maneuvered during VR gameplay by pedaling and steering their virtual character by leaning their bodies left and right. (Daniel et al., 2020).
  group (B) control group :Cycling by traditional stationary bike: Participants will require to continuously pedal using the pulse oximeter for HR monitor. Research personnel monitored participants during the session adjusting pedal-resistance to ensure that the participants stayed within their target HR zone. (Daniel et al., 2020).
  Other Names: group (B) control group : Cycling by traditional stationary bike:

SUMMARY:
Low levels of physical activity and sedentary lifestyle have become a major public health problem contributing to the prevalence of many chronic diseases and reduced life expectancy worldwide, and also increase the risk of heart disease, stroke, hypertension, type 2 diabetes, dementia, depression, excessive weight gain, and breast and colon cancer. Physical activity improves functional health and quality of life. (Iva Sklempe Kokic et al., 2019).

In Middle East, Insufficient physical activity and sedentary behavior are key risk factors for obesity and other diseases leading to premature mortality. Regular physical activity can improve self-esteem, cognitive performance, and academic achievement in young people. (Sonia Chaabane et al., 2020).

University students, due to the time spent in classes, studying or in front of computers, form part of the population most at risk of adopting sedentary behavior. Different studies have shown that the transition to university studies is usually associated to a decrease in physical activity and an increase in sedentary behavior as a result of lifestyle changes, as well as psychosocial factors. (Cotton et al., 2016).

Exercise is often perceived as boring and hard, thereby causing adults and students shy away from physical activity -related behaviors after long days of work and/or school. Instead, individuals are more interested in leisure activities, such as video games, Thus, the combination of video games and engaging in physical activity (e.g., virtual reality -integrated exercise) may

trigger their interest and improve their physical activity behavior. (Jiali Qian et al., 2020).

So, this trial aim to find if the virtual reality exercise as a new modality will make sedentary physical student more interest to adherent to exercise than conventional aerobic training so makes them more physically active which will enhance their academic performance and endurance.

DETAILED DESCRIPTION:
This study will design to compare the effect of Virtual Reality Exercise versus aerobic training on performance and endurance in physical therapy students.

I-Subjects:

This study will be carried out on sixty physical therapy students (female-class I obesity) will selected from faculty of physical therapy, all participants will be randomly assigned to two equal group in number, their ages will be ranged from (18-25) years.

Ethical consideration:

The purpose, nature and potential risks of the study will explain to participants. All participants will sign a consent form prior to participation in the study as shown in appendix I. no of approval…………

Inclusion criteria:

The subject selection will be according to the following criteria:

* Age between 18 and 25 years.
* Female only will participate in the study.
* Class I obesity, Body mass index is (30.0 to 34.9).
* No diseases/conditions preventing physical activity participation.

Exclusion criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Have any cardiovascular, cerebrovascular, or neurological diseases.
* Have any attention disorders or physical disability.
* Previously played the virtual reality exercise that will applied in this thesis.

The subjects participating in the study will be randomly assigned to two equal group in number:

- Group A (Study group): (Thirty participant) The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min

cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller).

- Group B (Control group): (Thirty participant) The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of cycling session by traditional stationary bike.

II-Materials:

1. Evaluation tools:

   1. Height/weight chart :

      To calculate body mass index, as shown in appendix II. ( Karoline Hood et al., 2019).
   2. pulse oximeter: To measure oxygen saturation and HR before and after each session. And monitor HR during session.

      (Digital Fingertip Pulse Oximeter LED Display Blood Oxygen and HR, Brand: CONTEC, Manufacturer Number: 2724295057898, made in china).
   3. The 6-min walk test (6MWT):

      participant is asked to walk as far as possible along a 30-m minimally trafficked corridor for a period of 6 min with the primary outcome measure being the 6-min walk distance (6MWD) measured in meters. (PriyaAgarwala et al ., 2020).
   4. Measure estimated vo2 max:

      At first Determine resting heart rate by pulse oximeter Then Calculate maximum heart rate by subtract age from 220. Then calculate estimated VO2 max by formula.
      * VO2 max = 15 x (HRmax/HRrest).
      * The units for VO2 max are milliliters of oxygen per kilogram of body weight per minute (mL/kg/min). (Davies et al., 2020).
   5. The McArdle step test OR Queens college step test (QCT):

      The participant steps up and down on the platform at a rate of 22 steps per minute for females. The participants are to step using a four-step cadence, 'up-up-down-down' for 3 minutes. The participant stops immediately on completion of the test, and the heart beats are counted for 15 seconds from 5-20 seconds of recovery. Multiply this 15 second reading by 4 will give the beats per minute (bpm) value to be used in the calculation below. an estimation of VO2max can be calculated from the test results, using this formula. A rating can be determined using the VO2max norms.

      women: VO2max(ml/kg/min) = 65.81 - (0.1847 x heart rate (bpm)) (Çağtay Maden et al., 2022).
   6. The Perceived Stress Scale (PSS):

      Participant ask to indicate how often he felt or thought during the last month. Ten questions for each question participant choose from the following alternatives: 0 - never 1 - almost never 2 - sometimes 3 - fairly often 4 - very often. as shown in appendix III (Miguel A. Vallejo et al., 2018).
   7. The Ardell Wellness Stress Test:

      In this scale participant ask to rate satisfaction with each of the following items: (0 = Indifferent, + 1 = Mildly happy, + 2 = Very happy, + 3 = Ecstatic, -1 = Mildly disappointed, - 2 = Very disappointed, - 3 = Completely dismayed). as shown in appendix IV (Daksh Sharma et al., 2018).
   8. Stress Coping Resources Inventory: A Self-Assessment:

   participant ask to answer questions relate to factors most closely associated with the capacity to cope successfully with stress. Participant ask to Circle the letter which lists the option that he choose and Answer each question as honestly as possible. A perfect score will be 4. as shown in appendix V (Jesús de la Fuente et al., 2018).
2. Therapeutic tools:

   1. Fully Immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller):

      (Oculus Quest virtual reality (VR) headset with hand controller and software using Unreal Engine 4.20, 3ds Max 2019, and Substance Designer 2018 software), made in Japan.
   2. Traditional stationary bike:

      Traditional stationary cycling will complete on a Spirit Fitness XBU55 Upright Bike (Spirit Fitness, Jonesboro, AR), made in china.

      III-Methods:

      The intervention will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up will precede each session and 10-min resting phase after each session with the actual time of each session is 30 minute. (Chao Lan et al., 2022).

      Participants will require to continuously pedal while maintaining an HR between 65% and 85% of their age predicted maximum HR-tracked using the HR monitor in pulse oximeter. (Daniel et al., 2020).

      The participants will divide into two group equal in number:

      Group A (Study group): (Thirty participant) The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller).

      - virtual reality cycling by fully immersive Head-Mounted Display virtual reality (Oculus Quest virtual reality (VR) headset with hand controller):

      The VR cycling session utilized the VZFIT VR Exercise Bike (VZFIT, Cambridge, MA), which syncs with the Sony PlayStation 4 and PlayStation VR headset (Sony, Tokyo, Japan) via integrated sensors. Participants who wore prescription glasses were allowed to wear their glasses during this session and a trained research assistant adjusted the VR headset comfortably over the glasses to ensure all participants had optimal vision during gameplay. The associated VZFIT Arcade Game suite houses numerous VR mini-games within which ''Race Car'' and ''Le Tour''-virtual racecar and cycling racing games, respectively-were selected for play. These games were selected as preliminary pilot trials indicated these games to be most intense. Players maneuvered during VR gameplay by pedaling and steering their virtual character by leaning their bodies left and right. (Daniel et al., 2020).
      * Group B (Control group): (Thirty participant) The program of treatment will be 3 times a week lasting for 8 weeks. A standardized 5- min warm-up phase will precede each session and 10-min cooling down phase after each session with the actual time of each session is 30 minute. 30 minutes of cycling session by traditional stationary bike.
      * Cycling by traditional stationary bike:

      Participants will require to continuously pedal using the pulse oximeter for HR monitor. Research personnel monitored participants during the session adjusting pedal-resistance to ensure that the participants stayed within their target HR zone. (Daniel et al., 2020).

      Statistical procedures:

      Statistical Package for Social Sciences (SPSS)

      Descriptive statistics:

      In this study, the descriptive statistics (the mean and the standard deviation) will be calculated for all subjects in the two groups of the study to determine the homogeneity of the groups.

      Analytical statistics:

      Comparison will make by student's t-test to compare the variables between the two groups of the study. Paired t-test will use to compare before and after treatment in the same group. A value of p<0.05 will be considered statistically significant (Prabhaker Mishra et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:
* Age between 18 and 25 years.
* Female only will participate in the study.
* Class I obesity, Body mass index is (30.0 to 34.9).
* No diseases/conditions preventing physical activity participation.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* Have any cardiovascular, cerebrovascular, or neurological diseases.
* Have any attention disorders or physical disability.
* Previously played the virtual reality exercise that will applied in this thesis.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological sex is a determinant of cardio respiratory endurance and performance: adult males are faster, stronger, more powerful than females because of fundamental sex differences in anatomy and physiology dictated by sex chromosomes.
Enrollment: 60 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The 6-min walk test (6MWT): | change in distance so change in cardio respiratory endurance before the intervention and after the intervinton (after 8 weeks)
  participant is asked to walk as far as possible along a 30-m minimally trafficked corridor for a period of 6 min with the primary outcome measure being the 6-min walk distance (6MWD) measured in meters. (PriyaAgarwala et al ., 2020).
Estimated vo2 max: | change in estimated vo2 max so change in cardio respiratory endurance before the intervention and after the intervinton (after 8 weeks)
  At first Determine resting heart rate by pulse oximeter Then Calculate maximum heart rate by subtract age from 220. Then calculate estimated VO2 max by formula.
  * VO2 max = 15 x (HRmax/HRrest).
  * The units for VO2 max are milliliters of oxygen per kilogram of body weight per minute (mL/kg/min). (Davies et al., 2020).
The McArdle step test OR Queens college step test (QCT): | change in Queens college step test (QCT) result so change in cardio respiratory endurance before the intervention and after the intervinton (after 8 weeks)
  The participant steps up and down on the platform at a rate of 22 steps per minute for females. The participants are to step using a four-step cadence, 'up-up-down-down' for 3 minutes. The participant stops immediately on completion of the test, and the heart beats are counted for 15 seconds from 5-20 seconds of recovery. Multiply this 15 second reading by 4 will give the beats per minute (bpm) value to be used in the calculation below. an estimation of VO2max can be calculated from the test results, using this formula. A rating can be determined using the VO2max norms.
  women: VO2max(ml/kg/min) = 65.81 - (0.1847 x heart rate (bpm)) (Çağtay Maden et al., 2022).
The Perceived Stress Scale (PSS): | change in performance or behaviour before the intrvention and after (8 weeks)
  Participant ask to indicate how often he felt or thought during the last month. Ten questions for each question participant choose from the following alternatives: 0 - never 1 - almost never 2 - sometimes 3 - fairly often 4 - very often. as shown in appendix III (Miguel A. Vallejo et al., 2018).
The Ardell Wellness Stress Test: | change in performance or behaviour before the intrvention and after (8 weeks)
  In this scale participant ask to rate satisfaction with each of the following items: (0 = Indifferent, + 1 = Mildly happy, + 2 = Very happy, + 3 = Ecstatic, -1 = Mildly disappointed, - 2 = Very disappointed, - 3 = Completely dismayed). as shown in appendix IV (Daksh Sharma et al., 2018).
Stress Coping Resources Inventory: A Self-Assesment scale: | change in performance or behaviour before the intrvention and after (8 weeks)
  participant ask to answer questions relate to factors most closely associated with the capacity to cope successfully with stress. Participant ask to Circle the letter which lists the option that he choose and Answer each question as honestly as possible. A perfect score will be 4. as shown in appendix V (Jesús de la Fuente et al., 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Hany Obeya, assistant professor, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Giza , Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No